CLINICAL TRIAL: NCT03900078
Title: Inzisionelle Negative Drucktherapie Nach Resektion Von Weichteiltumoren - Eine Prospektive, Randomisierte, Kontrollierte Klinische Studie
Brief Title: Incisional Negative Pressure Wound Therapy for Resection of Soft Tissue Tumors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ruhr University of Bochum (Other)
Responsible Party: Principal Investigator, Mehran Dadras, MD, Consultant, Department of Plastic Surgery, Ruhr University of Bochum
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18-6411-BR
Record Dates: First submitted 2019-03-26; First posted 2019-04-02 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Soft Tissue Sarcoma; Lipoma; Tumor
MeSH Terms: conditions — Sarcoma; Lipoma; Neoplasms | interventions — Bandages

STUDY DESIGN:
Intervention Model Description: RCT with two therapy arms.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): After subcuticular skin suture, patients receive standard dressing with adhesive wound tapes.
  Interventions: Other: Wound dressing with adhesive tapes
- Incisional negative pressure group (Experimental): After subcuticular skin suture, patients receive an incisional negative pressure dressing for 5 days.
  Interventions: Other: Incisional negative pressure wound therapy

INTERVENTIONS:
Other: Incisional negative pressure wound therapy — A negative pressure dressing is applied to the skin incision.
  Arms: Incisional negative pressure group
Other: Wound dressing with adhesive tapes — Regular adhesive wound tapes are applied over the closed skin.
  Arms: Control group

SUMMARY:
This study is aimed to examine the value of incisional negative pressure therapy after resection of soft tissue tumors. Its a prospective randomized trial comparing incisional negative pressure to standard wound dressings.

DETAILED DESCRIPTION:
Wound healing after resection of large soft tissue tumors is often impaired by large dead space and fluid collection, potentially resulting in seroma formation and infection. Aim of the study is to compare negative pressure wound therapy to standard wound dressing in terms of quantity of drainage fluid and wound healing complications.

ELIGIBILITY:
Inclusion Criteria:

* Soft tissue tumor of extremities or trunk with expected resection of >10cm tissue in any dimension.

Exclusion Criteria:

* No primary skin closure.
* Skin infection in area of operation (e.g. acne inversa).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2020-08-01 (Actual); Study Completion 2020-09-15 (Actual)

PRIMARY OUTCOMES:
Amount of drainage fluid | up to 14 days postoperatively
  Measurement of total fluid amounts in drains and negative pressure device

SECONDARY OUTCOMES:
Wound complications | 3 months
  Assessment of course of wound healing, necessary operative revisions, seroma formation
Wound margin perfusion | 5 days postoperatively
  Measurement with laser doppler

CONTACTS AND LOCATIONS:
Overall Officials: Björn Behr, MD, Principal Investigator — Berufsgenossenschaftliches Universitätsklinikum Bergmannsheil Bochum; Mehran Dadras, MD, Study Director — Berufsgenossenschaftliches Universitätsklinikum Bergmannsheil Bochum
Locations (1):
- Berufsgenossenschaftliches Universitätsklinikum Bergmannsheil, Bochum, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No